CLINICAL TRIAL: NCT06921967
Title: A Comparison of Ocular Health and Visual Quality With Corneal and Scleral Rigid Gas Permeable Lenses in Keratoconus Patients
Brief Title: Effect of Corneal and Scleral RGP Lenses on Ocular Health and Visual Quality in Keratoconus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2500206
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-03

CONDITIONS: Keratoconus; Irregular Astigmatism
Keywords: Contact Lenses; Scleral Lenses; Corneal Lenses; Rigid gas permeable lenses; Rigid lenses; GP lenses; RGP lenses; Visual Acuity; Contrast Sensitivity; Higher Order Aberrations; Dry Eye Disease; Irregular Astimatism; Keratoconus
MeSH Terms: conditions — Keratoconus; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Corneal Rigid Gas Permeable Contact Lens (Active Comparator): Small diameter RGP lens (TD < HVID).
  Interventions: Device: Rose K2
- Scleral Rigid Gas Permeable Contact Lens (Active Comparator): Large diameter RGP lens (TD>HVID).
  Interventions: Device: Onefit MED

INTERVENTIONS:
Device: Rose K2 — Corneal RGP lens with flexible parameters.
  Arms: Corneal Rigid Gas Permeable Contact Lens
Device: Onefit MED — Scleral RGP lens with flexible parameters.
  Arms: Scleral Rigid Gas Permeable Contact Lens

SUMMARY:
This study aims to compare the ocular health and visual quality of corneal rigid gas permeable lenses (CRGPL) and scleral rigid gas permeable lenses (SRGPL) for patients with keratoconus in a crossover clinical trial. The study will analyze subjective and objective outcomes, including best corrected visual acuity, contrast sensitivity, higher-order aberrations and subjective perception of visual function and comfort. It will also investigate the impact of both lens types on the health of the ocular surface, including evaluation of corneal, conjunctival, and scleral tissues, and tear film. Only one randomized controlled trial has compared the effect of CRGPL and SRGPL wear for patients with an ectatic corneal disorder. With the increasing popularity of SRGPL, examining the differences in efficacy, safety, and patient-reported outcomes between the two types of lenses is increasingly relevant.

DETAILED DESCRIPTION:
A comparison of ocular health and visual quality with corneal and scleral rigid gas permeable lenses in keratoconus patients

1. Introduction

1.1 Purpose: Keratoconus is an ocular disease, causing progressive thinning and steepening of the cornea, which results in irregular astigmatism and reduced visual quality. Irregular astigmatism induced by an irregular anterior cornea can effectively be corrected with rigid gas permeable (RGP) lenses. The purpose of this study is to compare subjective and objective outcomes from corneal rigid gas permeable lens (CRGPL) and scleral rigid gas permeable lens (SRGPL) wear in patients with keratoconus.

The following three aims will be pursued during a randomized clinical trial (RCT)

1. To compare the subjective perception of visual function (SPVF), subjective perception of comfort (SPC) and objective measures for visual quality, including best corrected visual acuity (BCVA) and contrast sensitivity (CS), between CRGPL and SRGPL wear, for patients diagnosed with keratoconus.
2. To analyze the effect of CRGPL and SRGPL on higher order aberrations (HOA) for patients with keratoconus.
3. To investigate the impact of CRGPL and SRGPL wear on the ocular surface, including analysis of the corneal, conjunctival, and scleral tissue, as well as tear film analysis, for patients with keratoconus.

1.2 Hypothesis

1. SPVF and SPC will be significantly better for SRGPL wear compared to CRGPL wear, but the difference in clinical findings for visual quality will be insignificant.
2. The difference in reduction of HOA between CRGPL and SRGPL wear will be insignificant, but the overall HOA for both interventions will decrease significantly compared to baseline.
3. Significant variation in health of the anterior eye will be observed for CRGPL and SRGPL wear. SRGPL wear will more frequently exhibit adverse effects at the conjunctival and scleral tissue, whereas the corneal tissue will show more complications with CRGPL wear. Symptoms and clinical findings related to dry eye disease (DED) will be significantly superior with SRGPL wear.

2. Background

2.1 RGP lenses Fitting RGP lenses for patients with an irregular cornea, such as keratoconus, is a common optical rehabilitating treatment. Due to elevated HOA in patients with keratoconus, RGP lenses have the distinct advantage of significantly improving the visual quality through a reduction in aberrations from the anterior cornea with the tear lens between the cornea and the lens. Both CRGPL and SRGPL wear have been shown to potentially delay the need for corneal transplants in patients with keratoconus.

A CRGPL is designed to fit within the corneal diameter whereas the SRGPL is produced in a larger diameter, and designed with a bearing that rests solely on the conjunctival tissue. CRGPL fitting for keratoconus has traditionally followed one of three different design objectives. Apical clearance, apical touch, or three-point touch. The three-point touch method has shown better fitting success compared to the apical touch, which has the added risk of potentially inducing corneal scarring. The SRGPL has the unique advantage of being fitted without having any contact with the irregular cornea of patients with keratoconus and is increasingly useful in more advanced cases.

The effect on visual quality from CRGPL and SRGPL wear on patients with an ectatic corneal disorder has been compared in only one RCT with a study population consisting of 34 patients successfully fitted with CRGPL. Patients were fitted with both CRGPL and SRGPL designs in a crossover study. The difference in BCVA and CS between the two lens types was not statistically significant. This study differs by analyzing a larger variety of parameters related to ocular health, the tear film and higher order aberrations. The study population is also expected to be more homogeneous, since it will consist solely of patients with keratoconus and with no prior history of RGP lens wear, to minimize the risk of bias.

2.2 Higher order aberrations The ocular structures responsible for the refractive properties of the eye are the cornea and the crystalline lens. The shape and regularity of these structures influence how much the wavefront will deviate from an ideal wavefront. This deviation is also known as wavefront aberration. Wavefront aberrations are commonly categorized as lower-order aberrations (LOA) or higher-order aberrations (HOA) and can be described using the Zernike polynomials. Some HOA explained through Zernike polynomials, such as coma and trefoil, are most often seen in irregular corneas, and are usually managed with RGP lenses. Wavefront aberrations are quantifiable using an aberrometer, making it possible to compare the effect of different lens designs on the amount of residual HOA.

2.3 Complications from RGP lens wear Contact lens wear, regardless of modality, will potentially cause complications. For CRGPL most complications are located at the cornea, palpebrae, and tear film. Complications from CRGPL wear include 3 and 9 o'clock corneal staining, mechanical corneal staining, and vascularized limbal keratitis. Studies have also shown a potential risk of developing ptosis from CRGPL wear.

SRGPL wear potentially induces corneal oedema and conjunctival prolapse. From multiple smaller studies patients with keratoconus, wearing a modern SRGPL, exhibited an average corneal oedema of ~2%. Blurred vision from tear reservoir debris has also been observed in patients wearing a SRGPL. This phenomenon is known as midday fogging and has been estimated to occur in about 26-46% of SRGPL wearers.

3. Materials and methods The study population will consist of patients with keratoconus referred to the Department of Ophthalmology at Aarhus University Hospital.

Suitable subjects will be invited to participate in the study, and randomized to start with one of two interventions, CRGPL or SRGPL wear in a crossover clinical trial. Study subjects must comply with the following inclusion criteria: Keratoconus, best spectacle corrected visual acuity >0.00 log of minimum angle of resolution (logMAR) and age between 18 to 40. The exclusion criteria for this study are: K-max >60D, RGP lens wear at baseline and ocular surface disease, verified through examination of the ocular surface and patient history.

The study involves analysis of multiple different outcomes but to determine an appropriate sample size, BCVA using logMAR has been chosen as the primary outcome and therefore the sample size is calculated per findings related to that.

The mean logMAR for patients with keratoconus wearing a CRGPL from the studies used is 0.08 (0.10), and 0.18 (0.17) for SRGPL wear. Sample size calculations with α = 0.05 and β = 0.90 yield a required study population of 35 subjects, to detect a difference of 0.10 logMAR. To account for potential drop-out this study will aim to include 50 subjects.

Aim 1: To investigate the visual quality of patients with keratoconus during both CRGPL and SRGPL wear, BCVA using ETDRS standard charts, translated to logMAR units, and CS measured with the Pelli Robson chart, will be obtained. Furthermore, the SPVF will be analyzed using the validated Visual Function Questionnaire (VEQ-25), translated to a Danish validated version. The SPC will be quantified with a questionnaire developed specifically for this study. For fitting of contact lenses, corneal shape will be measured with the Pentacam HR tomography (Oculus, Switzerland) device and the Heidelberg SPECTRALIS OCT device (Heidelberg Engineering, UK).

Aim 2: The effect of CRGPL and SRGPL on the amount of HOA during lens wear will be measured using Hartmann Shack aberrometry with the Visual Adaptive Optics simulator (VAO) (Voptica, Spain).

Aim 3: During this part of the study the ocular health will be monitored before, during, and after CRGPL and SRGPL wear. The ocular health examination will include standardized grading of conjunctival and limbal hyperaemia, corneal neovascularization, corneal oedema, and staining of the ocular surface. The examination will be quantified using the Efron Grading scale, and documented with slit lamp photography. Corneal epithelial thickness and corneal tomography will also be examined before and after each intervention. Symptoms and clinical findings related to dry eye disease (DED) will be evaluated using the validated symptom survey "Ocular Surface Disease Index" (OSDI), translated to Danish and measured with break-up time (BUT).

4. Ethical considerations Since contact lenses are classified as medical devices, approval has been obtained from the Danish Medical Research Ethics Committees. When patients are invited to participate in the study, they will receive written information on the purpose of the study including an explanation of risks and benefits of the interventions. To participate an informed consent form must be obtained. The study will be conducted in agreement with the declaration of Helsinki, and patient data will be stored in agreement with the relevant Danish law. Since the intervention is to be administered and cared for by the patients at their residence, proper instruction of use will be delivered both in writing and verbally in the clinic.

5. Perspectives The prevalence of keratoconus shows substantial variation globally, with epidemiological studies estimating it between 0.2 and 4,790 per 100,000 persons. In Denmark the prevalence was estimated, by Bak-Nielsen et al (2019), to 40 per 100,000 persons. Research indicate that the incidence of patients with keratoconus has increased significantly in Denmark over the last 30 years. Nielsen et al (2007) estimated the incidence to 1.3 per 100,000 person-year based on data from 1995 to 2005. Bak-Nielsen et al (2019) estimated the same incidence to 3.8 per 100,000 person-year based on data from 2011 to 2015. The authors attribute a large portion of the increase in incidence to the introduction of CXL, which has changed the referral pattern. Treatment with CXL reduce the need for corneal transplantation, improves visual quality and reduces cone progression. Patients with keratoconus post CXL, generally still require RGP lenses as they remain the best option for improving visual quality.

The "International Contact Lens Prescribing"-reports investigate global contact lens prescribing trends. In 2013 scleral lens fits accounted for ~6% of all RGP lens fits reported, that increased to 22% in 2023. In Denmark there is a reported increase in RGP lens fits of total lens fits. In 2013 RGP lens fits accounted for 8% of all lens fits reported, this increased to 18% in 2023. With the increasing popularity of scleral lenses and the growing number of RGP lens fits reported in Denmark, research examining the differences in efficacy, safety and patient reported outcomes between the two types of lenses are increasingly relevant.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus, best spectacle corrected visual acuity >0.00 log of minimum angle of resolution (logMAR) and age between 18 to 40

Exclusion Criteria:

* K-max >60D, RGP lens wear at baseline and ocular surface disease, verified through examination of the ocular surface and patient history

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 6 weeks with each intervention. 13 weeks total, incl. 1 week washout.
  Comparison of Best Corrected Visual Acuity, with the two interventions, at the end of 6 weeks of lens wear. Measured with ETDRS charts, converted to logMAR units.

SECONDARY OUTCOMES:
Contrast Sensitivity | 6 weeks with each intervention. 13 weeks total, incl. 1 week washout.
  Comparision of contrast sensitivity with the two interventions, measured with a Pelli Robson Chart.
Higher Order Aberrations (HOA) | 6 weeks with each intervention. 13 weeks total, incl. 1 week washout.
  Comparison of HOA with the two interventions at the end of 6 weeks of lens wear. Measured with the Visual Adaptive Optics Simulator by Voptica. Root Mean Square value in microns.
Tear break-up time (TBUT) | 6 weeks with each intervention. 13 weeks total, incl. 1 week washout.
  Comparison of Tear break-up time with the two interventions at the end of 6 weeks of lens wear. Using fluorescein and slit lamp to capture the break-up time in seconds.
Anterior ocular health markers | 6 weeks with each intervention. 13 weeks total, incl. 1 week washout.
  Comparison of anterior ocular health with the two interventions at the end of 6 weeks of lens wear. Using fluorescein and slit lamp to grade with the Efron Grading Scale. Scored on a scale from 0 to 4 with higher values representing worse outcomes.
Corneal Epithelial Thickness | 6 weeks with each intervention. 13 weeks total, incl. 1 week washout.
  Comparison of the corneal epithelial thickness with the two interventions at the end of 6 weeks of lens wear. Using Pentacam HR from Oculus.
Corneal Tomography | 6 weeks with each intervention. 13 weeks total, incl. 1 week washout.
  Comparison of the corneal tomography with the two interventions at the end of 6 weeks of lens wear. Using Pentacam HR from Oculus.
Subjective Perception of Comfort (SPC) | 6 weeks with each intervention. 13 weeks total, incl. 1 week washout.
  Comparison of the SPC with the two interventions at the end of 6 weeks of lens wear. Quantified with a survey developed for this study. Minimum score 8 maximum 40, higher values indicate better comfort.
Subjective Percepton of Visual Function (SPVF) | 6 weeks with each intervention. 13 weeks total, incl. 1 week washout.
  Comparison of the SPVF with the two interventions at the end of 6 weeks of lens wear. Quantified with the validated Danish translation of the VEQ-25 survey. Scored on a scale from 0 to 100, higher values indicate better functioning.
Dry Eye Symptoms | 6 weeks with each intervention. 13 weeks total, incl. 1 week washout.
  Comparison of Dry Eye Symptoms with the two interventions at the end of 6 weeks of lens wear. Quantified with a Danish translation of the validated symptom survey Ocular Surface Disease Index (OSDI). Scored on a scale of 0 to 100, with higher values representing greater disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morgan P, Woods C, Tranoudis I, Efron N, Jones L, Faccia P, et al. International Contact Lens Prescribing in 2023. CONTACT LENS SPECTRUM. 2024;39:20-2,4,6-8
- [Background] Morgan P, Woods C, Tranoudis I, Helland M, N E, M T, et al. International Contact Lens Prescribing in 2013. Contact Lens Spectrum. 2014;29:30-5
- [Background] Mandathara PS, Kalaiselvan P, Rathi VM, Murthy SI, Taneja M, Sangwan VS. Contact lens fitting after corneal collagen cross-linking. Oman J Ophthalmol. 2019 Oct 11;12(3):177-180. doi: 10.4103/ojo.OJO_43_2018. eCollection 2019 Sep-Dec. PMID 31902993
- [Background] Nielsen K, Hjortdal J, Aagaard Nohr E, Ehlers N. Incidence and prevalence of keratoconus in Denmark. Acta Ophthalmol Scand. 2007 Dec;85(8):890-2. doi: 10.1111/j.1600-0420.2007.00981.x. Epub 2007 Jul 23. PMID 17645421
- [Background] Bak-Nielsen S, Ramlau-Hansen CH, Ivarsen A, Plana-Ripoll O, Hjortdal J. Incidence and prevalence of keratoconus in Denmark - an update. Acta Ophthalmol. 2019 Dec;97(8):752-755. doi: 10.1111/aos.14082. Epub 2019 Apr 9. PMID 30964230
- [Background] Ozcura F, Aydin S, Helvaci MR. Ocular surface disease index for the diagnosis of dry eye syndrome. Ocul Immunol Inflamm. 2007 Sep-Oct;15(5):389-93. doi: 10.1080/09273940701486803. PMID 17972223
- [Background] Efron N, Morgan PB, Katsara SS. Validation of grading scales for contact lens complications. Ophthalmic Physiol Opt. 2001 Jan;21(1):17-29. PMID 11220037
- [Background] Sorensen MS, Andersen S, Henningsen GO, Larsen CT, Sorensen TL. Danish version of Visual Function Questionnaire-25 and its use in age-related macular degeneration. Dan Med Bull. 2011 Jun;58(6):A4290. PMID 21651879
- [Background] Barnett M, Courey C, Fadel D, Lee K, Michaud L, Montani G, van der Worp E, Vincent SJ, Walker M, Bilkhu P, Morgan PB. CLEAR - Scleral lenses. Cont Lens Anterior Eye. 2021 Apr;44(2):270-288. doi: 10.1016/j.clae.2021.02.001. Epub 2021 Mar 25. PMID 33775380
- [Background] Hwang K, Kim JH. The Risk of Blepharoptosis in Contact Lens Wearers. J Craniofac Surg. 2015 Jul;26(5):e373-4. doi: 10.1097/SCS.0000000000001876. PMID 26102541
- [Background] Efron N. Contact Lens Practice. 4th ed. New Dehli: Elsevier; 2023
- [Background] Rosenfield M, Logan N. Optometry : science, techniques and clinical management. 2nd ed. Edinburgh: Butterworth Heinemann Elsevier; 2009
- [Background] Levit A, Benwell M, Evans BJW. Randomised controlled trial of corneal vs. scleral rigid gas permeable contact lenses for keratoconus and other ectatic corneal disorders. Cont Lens Anterior Eye. 2020 Dec;43(6):543-552. doi: 10.1016/j.clae.2019.12.007. Epub 2020 Jan 8. PMID 31924530
- [Background] Romero-Jimenez M, Santodomingo-Rubido J, Gonzalez-Meijome JM. An assessment of the optimal lens fit rate in keratoconus subjects using three-point-touch and apical touch fitting approaches with the rose K2 lens. Eye Contact Lens. 2013 Jul;39(4):269-72. doi: 10.1097/ICL.0b013e318295b4f4. PMID 23771007
- [Background] Michaud L, Lipson M, Kramer E, Walker M. The official guide to scleral lens terminology. Cont Lens Anterior Eye. 2020 Dec;43(6):529-534. doi: 10.1016/j.clae.2019.09.006. Epub 2019 Sep 25. PMID 31561849
- [Background] Ling JJ, Mian SI, Stein JD, Rahman M, Poliskey J, Woodward MA. Impact of Scleral Contact Lens Use on the Rate of Corneal Transplantation for Keratoconus. Cornea. 2021 Jan;40(1):39-42. doi: 10.1097/ICO.0000000000002388. PMID 32452985
- [Background] Koppen C, Kreps EO, Anthonissen L, Van Hoey M, Dhubhghaill SN, Vermeulen L. Scleral Lenses Reduce the Need for Corneal Transplants in Severe Keratoconus. Am J Ophthalmol. 2018 Jan;185:43-47. doi: 10.1016/j.ajo.2017.10.022. Epub 2017 Nov 16. PMID 29103959
- [Background] Santodomingo-Rubido J, Carracedo G, Suzaki A, Villa-Collar C, Vincent SJ, Wolffsohn JS. Keratoconus: An updated review. Cont Lens Anterior Eye. 2022 Jun;45(3):101559. doi: 10.1016/j.clae.2021.101559. Epub 2022 Jan 4. PMID 34991971